CLINICAL TRIAL: NCT00626418
Title: A Single-blind, Placebo Controlled Sleep Laboratory Study of the Acute Effects of Aplindore in Restless Legs Syndrome
Brief Title: The Effects of Aplindore on the Treatment of Signs and Symptoms of Restless Legs Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Aplindore-101
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — aplindore fumarate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): This will be a crossover study. Ascending doses of active drug will be administered on study nights 3-5 with an option of 3 additional nights in an attempt to identify a tolerable efficacious dose. Night 1 will be an adaptation night and night two will be a placebo night.
  Interventions: Drug: Placebo
- 2 (Active Comparator): This will be a crossover study. Ascending doses of active drug will be administered on study nights 3-5 with an option of 3 additional nights in an attempt to identify a tolerable efficacious dose. Night 1 will be an adaptation night and night two will be a placebo night.
  Interventions: Drug: Aplindore

INTERVENTIONS:
Drug: Aplindore — Tablets 0.05, 0.1, 0.2, 0.3, 0.5 and 0.7 mg QD for up to 6 nights
  Arms: 2
Drug: Placebo — Placebo tablets
  Arms: 1

SUMMARY:
The purpose of this study is to assess the efficacy and tolerability of single doses of aplindore compared to placebo in RLS. Patients will be required to spend 5-8 nights in a sleep laboratory. This includes 1 adaptation night, 1 placebo night, and 3-6 drug treatment nights. Ascending doses of active drug will be administered on study nights 3 through 5 to determine the maximum well tolerated efficacious dose (defined as a decrease in Periodic Limb Movement Index (PLMI) of at least 50% from placebo baseline). If an efficacious dose cannot be identified the Investigator in consultation with the sponsor may decide to examine higher doses in up to 3 additional PSG nights in an attempt to identify a tolerable efficacious dose. This study will utilize up to 24 evaluable patients, each meeting International Classification of Sleep Disorders (ICSD-2) diagnostic criteria for primary RLS who are not currently taking any RLS medication including DAs ( and L-dopa) or who are able to discontinue their RLS medication at least 5 half-lives prior to the adaptation night.

DETAILED DESCRIPTION:
Restless legs syndrome (RLS) is a neurosensorimotor disorder of uncertain etiology that commonly disturbs sleep. The main feature of the disorder is paresthesia felt deep in the limbs that troubles the individual when he or she is at rest. The paresthesias of RLS commonly increase during the evening or the early part of the night. Patients are commonly less bothered by symptoms in the morning, unless they are severely affected. The repetitive movements that lead to arousal may also cause a subset of patients to become quite sleepy during the daytime. This sleepiness is usually not as severe as that found in patients with sleep apnea or narcolepsy but can be quite disruptive to quality of life and daytime functioning. Recent surveys indicate that RLS occurs in 10% to 15% of the North American population.

A common associated feature of RLS is Periodic Limb Movements during Sleep (PLMS). These are repetitive movements that typically occur as flexions of the foot, knee, and hip at intervals of 5 to 90 seconds. Most commonly, the interval is 20 to 40 seconds. The movements are present during non-rapid-eye-movement (REM) sleep and are less common during REM sleep. Population-based studies have found that RLS is associated with an increased risk for hypertension and coronary artery disease. Periodic leg movements -related repetitive nocturnal blood pressure fluctuations may contribute to this increased risk of cardiovascular disease especially in the elderly19. There is a possibility that dopamine agonist (DA) reduction of PLMS may mitigate the risk of the cardiovascular complications of RLS. The potential role of aplindore in reducing PLMS and nocturnal blood pressure fluctuations will be evaluated in this study.

Dopaminergic agents have become the most common medications used in the treatment of RLS and PLMS. Aplindore is an orally available, small molecule partial agonist of the D2 dopamine receptor. Preclinical in vitro and in vivo results have demonstrated the functional agonist selectivity of aplindore for supersensitive D2 receptors in the striatum, but not extra-striatal D2 receptors. Stimulation of D2 receptors in areas deficient in dopamine is attributed to aplindore's low intrinsic activity and high affinity for these receptors. Aplindore has been studied in preclinical toxicology studies in rats for up to 6 months and in monkeys for up to 1 year with safety margins in excess of 100-fold relative to projected human efficacious doses. The primary objective of this study is to assess the efficacy and tolerability of single doses of aplindore compared to placebo in RLS. The secondary objectives are to generate safety data with aplindore to support outpatient trials in RLS. b) To generate pilot data on the effects of aplindore on changes in blood pressure and heart rate associated with PLMS in patients with RLS. c) To understand the concentration-effect relationships of aplindore on RLS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Diagnosis of primary Restless Legs Syndrome (RLS) using ICSD-2 criteria:
* The patient reports an urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs.
* The urge to move or the unpleasant sensations begin or worsen during periods of rest or inactivity such as lying or sitting.
* The urge to move or the unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues.
* The urge to move or the unpleasant sensations are worse, or only occur, in the evening or night.
* The condition is not better explained by another current sleep disorder, medical or neurological disorder, mental disorder, medication use, or substance use disorder.
* International Restless Leg Syndrome Study Group (IRLSSG) RLS rating scale score > 15 at screening
* PLMI of greater than 10 per hour of total sleep time (TST) determined by PSG during the adaptation night;
* Body mass index (BMI) ≤ 35 kg/m2;
* In good general health as determined by a thorough medical history and physical examination (including vital signs), 12-lead ECG (lab tests mentioned below)
* Patients have clinical laboratory values within normal reference range or must not be clinically significantly abnormal as judged by the Investigator and approved by the Sponsor;
* Patients must be off all prescription drug therapy or OTC medication they may be taking for RLS as well as any other psychotropic medication for at least 5 half lives prior to adaptation night and off any investigational drug for at least 30 days;
* Patients taking prescription or over-the-counter medication for chronic medical conditions must be on stable doses of these medications for at least two weeks prior to participation in the study.
* If the patient is a female of childbearing potential, she must be using an acceptable method of contraception, must have a negative urine pregnancy test at screening, and must have a negative urine pregnancy test at the adaptation night. Acceptable methods of contraception are oral, intrauterine, implantable, injectable contraceptives or double barrier methods. After screening, patients using oral contraceptives must agree to add the double barrier method until 30 days following the last dose of study medication. Women on oral contraceptives must have been using them for at least one month prior to screening.
* Be able to read, understand, and provide written/dated informed consent before enrolling in the study, and must be willing to comply with all study procedures;
* Patients must be willing and able to be confined to the clinical research site for a period of 5 nights or more as required by the protocol.
* Patients must refrain from strenuous physical activity on the day of admission and on PSG days.

Exclusion Criteria:

* Clinically significant unstable medical illness;
* Evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease;
* History of non-Basal Cell cancer within 5 years of screening;
* History of non-gestational diabetes within 5 years of screening;
* A supine blood pressure > 140/90 mm/Hg at screening or adaptation;
* Clinically significant psychiatric illness, including chronic psychiatric illness or the history or presence of any Axis I condition;
* History or presence of chronic pain other than that associated with RLS;
* History of epilepsy or serious head injury;
* Clinically significant sleep apnea, narcolepsy, parasomnia as an adult, circadian rhythm disorder, or secondary causes of RLS;
* An apnea-hypopnea index (AHI) > 10, as assessed by PSG during the adaptation night
* Any condition that may affect oral drug absorption;
* Travel across more than three time zones, an expected change in sleep schedules of 6 hours or more, or involvement in night shift work within seven days prior to screening or during the study period;
* Any clinically significant abnormal finding on physical examination, vital signs, ECG, or clinical laboratory tests, as determined by the Investigator. (The QTcB interval must be ≤ 450 msec for males and ≤ 470 msec for females);
* History of allergies, or known sensitivity, hypersensitivity, or adverse reaction to any drug similar to aplindore;
* Pregnant or lactating females;
* Recent history (≤ one year) of alcohol or drug abuse, or current evidence of substance dependence or abuse as defined by DSM-IV criteria;
* Regular consumption of large amounts of xanthine-containing substances (i.e. more than 5 cups of coffee or equivalent amounts of xanthine-containing substances per day);
* Self report of the usual consumption of more than 14 units of alcohol per week;
* Secondary causes of RLS which will be ruled out by physical exam, medical history and clinical chemistries, including serum ferritin;
* Use of any investigational drug within 30 days prior to screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and tolerability of single doses of aplindore compared to placebo in RLS. | 5-8 Days

SECONDARY OUTCOMES:
To generate safety data with aplindore, to generate pilot data on the effects of aplindore on changes in blood pressure and heart rate associated with PLMS in patients with RLS, to understand the PK of aplindore. | 5-8 Days

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - MD Clinical, Hallandale, Florida
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Community Research, Crestview Hills, Kentucky
  - Clinilabs, Inc., New York, New York
  - Lynn Health Science Institute, Oklahoma City, Oklahoma